CLINICAL TRIAL: NCT01577329
Title: Mindfulness Mediation Intervention in COPD
Brief Title: Mindfulness Mediation Intervention in Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Roxane Raffin Chan, RN, PhD, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: um-nursing-meditation
Record Dates: First submitted 2012-04-11; First posted 2012-04-13 (Estimated); Results first posted 2017-08-02 (Actual); Last update posted 2017-08-02 (Actual); Status verified 2017-04

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: meditation; Chronic Obstructive Pulmonary Disease; Mindfulness; Anxiety; Breathing Patterns
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Anxiety Disorders | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- mindfulness meditation class (Experimental): Group class on mindfulness meditation. One hour weekly class led by nurse expert on meditation that includes mindfulness skills, body awareness skills and emotional awareness skills. Homework is assigned.
  Interventions: Behavioral: Mindfulness meditation
- wait list (No Intervention): Subjects assigned to the control group will continue with medical treatment as usual and be allowed to attend the mindfulness meditation class after week eight.

INTERVENTIONS:
Behavioral: Mindfulness meditation — Group class on mindfulness meditation. One hour weekly class led by nurse expert on meditation that includes mindfulness skills, body awareness skills and emotional awareness skills. Homework is assigned.
  Arms: mindfulness meditation class

SUMMARY:
The purpose of this study is to assess the feasibility and potential impact of an eight week program of meditation on expiratory time, anxiety and dyspnea in people with COPD.

DETAILED DESCRIPTION:
Chronic Obstructive Pulmonary Disease is a progressive multi-dimensional disease with a complex network of somatic and affective components. Anxiety is a common experience for persons with COPD both as a reaction to dyspnea (48) and as a separate co-morbid condition (10, 26). The presence of anxiety magnifies COPD symptoms and further impairs physical functioning (53). Both anxiety and COPD alter breathing patterns similarly causing irregular rapid shallow breathing at rest, which is inefficient and cannot adequately respond to increases in ventilatory demands from physical or emotional activity (121). Both COPD and anxiety are also associated with changes in neurological functioning. Whereas anxiety tends to be associated with increased amygdala activity (54), COPD is associated with a decrease in frontal cortex functioning (25, 28, 122). Persons with COPD who experience anxiety are less able to correctly process the level of physical and emotional demand for any given situation and their ability to meet that demand (46, 123). Pulmonary rehabilitation addresses both the physical and emotional symptoms of COPD, however gains in function are quickly lost over time (4). Evidence suggests that mindfulness based meditation can alter neural pathways to facilitate processing of emotions and increase quality of life for persons with COPD. The overall objective of this study is to assess the ability of persons with COPD to participate in a mindfulness meditation intervention and to examine the impact of mindfulness meditation on their anxiety levels and global sense of coherence. A modified version of Antonovsky's sense of coherence model will be used as the framework for this study. We will address the specific aims: 1) to determine the effects of mindfulness meditation on breathing patterns; 2) To determine the effects of mindfulness meditation on anxiety levels; 3) To determine self-reported adherence rates following an eight-week small group instructional course on mindfulness meditation, and 4) To determine the effects of mindfulness meditation on global sense of coherence levels in persons with COPD. The National Center for Complementary and Alternative Medicine identifies meditation as a form of CAM that focuses on the interaction among the brain, body, mind and behavior that is already practiced by 8% of persons who participate in CAM therapy. Meditation is rated a special priority research area by NCCAM.

ELIGIBILITY:
Inclusion Criteria:

* Any stage of Chronic Obstructive Pulmonary Disease
* Able to read and write English

Exclusion Criteria:

* Severe mental disability
* Inability to attend

Ages: 40 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2011-10; Primary Completion 2013-05 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roxane R Chan, RN, PhD (c), Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Chan RR, Giardino N, Larson JL. A pilot study: mindfulness meditation intervention in COPD. Int J Chron Obstruct Pulmon Dis. 2015 Mar 2;10:445-54. doi: 10.2147/COPD.S73864. eCollection 2015. PMID 25767382

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Change was made to original number of participants due to human error. 51 persons were approached regarding possible enrollment.
Period: Overall Study
Arm/Group | Mindfulness Meditation Class | Wait List
Started | 19 | 22
Completed | 16 | 22
Not Completed | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Meditation Class | Wait List | Total
Number analyzed (Participants) | 19 | 22 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 1 | 4
  >=65 years | 16 | 21 | 37
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.3 (5.2) | 68.7 (4.8) | 69.5 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 6 | 8 | 14
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 22 | 41

OUTCOME MEASURES:

1. Primary Outcome: Changes in Respiratory Rate
Description: Breathing patterns will be measured at baseline using inductive plethysmography at baseline and at week eight. During that eight week time period the treatment group will have been exposed to a once a week mindfulness meditation class and the control group will have been exposed to health care as usual.
Time Frame: baseline and at week eight
Measure: Mean (Standard Deviation); unit: Breaths per minute
Arm/Group | Mindfulness Meditation Class | Wait List
Number analyzed (Participants) | 16 | 22
Breaths per minute
  Baseline | 15.93 (2.82) | 17.18 (6.44)
  Follow-up | 21.31 (3.05) | 18.73 (4.31)
Statistical Analysis 1: Comparison: Mindfulness Meditation Class vs Wait List; This is a calculated P value comparing two groups at baseline and follow-up; Test type: Superiority or Other; p = 0.05, ANOVA — This is a calculated P value and was not adjusted for multiple comparisons

ADVERSE EVENTS:
Time Frame: Eight weeks
Arm/Group | Mindfulness Meditation Class | Wait List
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/19 | 0/22
Other Adverse Events (participants affected / at risk) | 0/19 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes